CLINICAL TRIAL: NCT06060028
Title: The Power of Touch. Randomized,Double-blind, Sham-controlled Crossover Trial of Interoceptive Non-invasive Tactile Stimulation for the Treatment of Osteoarthritis Chronic Associated Pain
Brief Title: The Power of Touch. Non-Invasive C-Tactile Stimulation for Chronic Osteoarthritis Pain
Acronym: TouchStim
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Auxologico Italiano (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 39A101
Record Dates: First submitted 2023-09-07; First posted 2023-09-29 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- General Practitioner (GP) care plus interoceptive non-invasive tactile stimulation treatment (Experimental): Participants will receive General Practitioner (GP) care and interoceptive non-invasive tactile stimulation (affective touch) for 30 min two times a week for 12 weeks.
  Interventions: Device: Interoceptive stimulation treatment with mechanical stimulation of C-LTMRs afferences
- GP care plus sham treatment (Sham Comparator): Participants will receive General Practitioner (GP) care and a sham stimulation for 30 min two times a week for 12 weeks.
  Interventions: Device: Sham treatment

INTERVENTIONS:
Device: Interoceptive stimulation treatment with mechanical stimulation of C-LTMRs afferences — The intervention is a non-invasive interoceptive stimulation (affective touch) delivered to the left volar forearm. The stimulation is delivered using a device with a small tactile probe that touches the skin in a circular motion. The device is designed to induce maximum firing frequency in the peripheral C-Ts nervous afferents, which respond to low-force, low-velocity stimuli, specifically 3 cm/sec, 2.5mN. The stimulation will be delivered in 18 blocks, each consisting of 6 short periods of stimulation of varying durations presented in random order, with pauses of 6 seconds after every single stimulation, the entire stimulation protocol will have a total duration of 30 minutes.
  Arms: General Practitioner (GP) care plus interoceptive non-invasive tactile stimulation treatment
Device: Sham treatment — In the sham condition, patients will receive a similar stimulation with the interoceptive tactile device, however, the device will be turned on for only 3 seconds every minute, and consequently turned off for 57 seconds. The entire duration of the stimulation will be approximately 30 minutes, similar to the experimental condition.
  Arms: GP care plus sham treatment

SUMMARY:
Osteoarthritis (OA) is a degenerative disease with a prevalence of up to 30% among adults over 45 years old. Moreover, elderly people over 60 years are more prone to develop a chronification of pain symptomatology. Chronic pain in OA enormously restricts patients' ability to perform their daily activities, eliciting psychological distress and mood alterations, and producing massive socioeconomic consequences. For these reasons, any non-invasive drug-free treatment that decreases chronic pain in OA requires serious evaluation.

This study aims to investigate the effectiveness of noninvasive interoceptive stimulation (affective touch) in treating chronic pain associated with osteoarthritis (OA).

This study aims to investigate the effectiveness of noninvasive interoceptive stimulation (affective touch) in treating chronic pain associated with osteoarthritis (OA).

DETAILED DESCRIPTION:
The current study aims to assess the long-term analgesic efficacy of interoceptive tactile stimulation in patients suffering from chronic moderate-to-severe osteoarthritis (OA) pain. The study will be a randomized, double-blind, sham-controlled crossover trial involving 60 OA patients with moderate-to-severe chronic pain. Patients will be randomly assigned to the treatment or control group and received interoceptive (affective touch) or control stimulation two days a week for 12 weeks. Patient will then undergo to a 4-week washout period, after that they will be assigned to the crossover treatment for another 12 weeks. The study will measure changes in pain and physical function, heart rate variability, as well as inflammatory and anti-inflammatory cytokines and medication intake, assessed at baseline, and at the end of each crossover phase. Follow-up measures will be assessed 4 weeks after the end of each crossover phase. Intermediate outcomes for pain and physical function, heart rate variability and medication intake will also be assessed after 4 and 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* osteoarthritis patients
* Age 45-90
* Diagnosis of OA ACR criteria
* Moderate-to-severe OA chronic pain.

Exclusion Criteria:

* other joint diseases
* trauma, or pain condition
* fibromyalgia
* BMI>39 kg/m2.

Ages: 45 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-07-06 (Actual); Primary Completion 2025-04-09 (Actual); Study Completion 2025-05-07 (Actual)

PRIMARY OUTCOMES:
the pain subscale scores from Western Ontario and McMaster Universities OA Index (WOMAC) | the change from baseline to week 12 in the pain subscale scores of the WOMAC
  A higher WOMAC score represented worse symptom severity. Measures are assessed in a modified intention-to treat population for all participants randomly assigned to groups and who attended a baseline visit.
the physical function subscale scores of the Western Ontario and McMaster Universities OA Index (WOMAC) | Will be the change from baseline to week 12 in the physical function subscale scores of the Western Ontario and McMaster Universities OA Index (WOMAC).
  A higher WOMAC score represented worse symptom severity. Measures are assessed in a modified intention-to treat population for all participants randomly assigned to groups and who attended a baseline visit.
the patient global assessment (PGA) of osteoarthritis. | Will be the change from baseline to week 12 in the patient global assessment (PGA)
  Measures are assessed in a modified intention-to treat population for all participants randomly assigned to groups and who attended a baseline visit.

SECONDARY OUTCOMES:
Long term changes of inflammatory cytokine plasmatic levels | the change from baseline to week 12
  Interleukin-10 (IL-10), Tumor necrosis factor alpha or TNF-α, interleukin 1 family of cytokine, IL-1β, Interleukin-6 (IL-6), Interleukin-4 (IL4)
Long term changes of stress/pain/anxiety-related hormone plasmatic levels cortisol and oxytocin | the change from baseline to week 12
  IL-10 and IL-4

OTHER OUTCOMES:
joint pain scores | the change pre-intervention and immediately after the intervention
  Pain Numeric Rating Scale (NRS). Minimum score 0 (no pain); maximum score 10 (worst pain imaginable). The higher the score the higher the pain.
rescue analgesic medication intake | the change from baseline to week 12
  change of amount of rescue analgesic medication intake (the lower the better)
change in sympathetic activity | the change pre-intervention and immediately after the intervention
  change in sympathetic activity (Low-Frequency power band index)
Short term changes of inflammatory cytokine and hormone plasmatic levels | the change pre-intervention and immediately after the intervention
  Interleukin-10 (IL-10), Tumor necrosis factor alpha or TNF-α, interleukin 1 family of cytokine or IL-1β, Interleukin-6(IL-6),Interleukin-4 (IL4), cortisol and oxytocin
the percentage of patients who responded to Western Ontario and McMaster Universities (WOMAC) | changes at week 12
  the percentage of patients who responded to treatment according to ≥30% and ≥50% changes at week 12 in the WOMAC pain and physical function subscale scores.
pain diary | two days a week in the 48 hours preceding the treatment sessions
  Pain weekly measures will be collected with a pain diary two days a week. In the dairy, patients will report pain ratings on the WOMAC pain subscale, to keep track of sudden variations in the symptomatology (i.e., flares) in the 48 hours preceding the treatment sessions.
change in parasympathetic activity | the change pre-intervention and immediately after the intervention
  change in parasympathetic activity (rMSSD index)
change in parasympathetic | the change pre-intervention and immediately after the intervention
  change in parasympathetic (HighFrequency power band index)

CONTACTS AND LOCATIONS:
Overall Officials: Daniele Di Lernia, Principal Investigator — Catholic University of the Sacred Heart of Milan
Locations (1):
- Cosimo Tuena, Milan, Lombardy, Italy